CLINICAL TRIAL: NCT00768417
Title: Mastication of Almonds: Effects of Lipid Bioaccessibility, Appetite, and Hormone Response
Brief Title: Availability of Lipids in Almonds in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Foods and Nutrition, Purdue University
Other Study IDs: 0511003189
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Obesity; Overweight
Keywords: Nuts; Lipids; Mastication; Bioaccessibility; Satiety; Hormones; Human
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, feces
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Participants: Participants completed all 3-arms of this cross-over design study.
  Interventions: Behavioral: 10 chews; Behavioral: 25 Chews; Behavioral: 40 Chews

INTERVENTIONS:
Behavioral: 10 chews — Participants were required to chew 55g grams of almonds per day for four days in 11, 5 gram portions. Almonds were to be chewed 10 times before swallowing.
  Other Names: Almonds
Behavioral: 25 Chews — Participants were required to chew 55g grams of almonds per day for four days in 11, 5 gram portions. Almonds were to be chewed 25 times before swallowing.
  Other Names: Almonds
Behavioral: 40 Chews — Participants were required to chew 55g grams of almonds per day for four days in 11, 5 gram portions. Almonds were to be chewed 40 times before swallowing.
  Other Names: Almonds

SUMMARY:
Evidence indicates that almond consumption is associated with multiple health benefits. However, nuts are commonly excluded from diets on the basis that their high energy content may induce weight gain. Evidence from numerous studies show that this is not the case, yet the mechanism responsible for the less than predicted effect on weight is unknown. This study aimed to examine the effects of increased mastication on lipid bioavailability and satiety related peptide released in humans. Its purpose is to provide valuable mechanistic data to support the results from previous completed clinical studies.

DETAILED DESCRIPTION:
This cross-over study consisted of three study periods of four consecutive days separated by at least one week. During each day of the three study periods, participants were required to consume 55g of almonds split up into 5 g portions. They were required to chew the almonds 10, 25, or 40 times before swallowing, depending on the treatment. During each treatment period, all participants followed the same procedures over the four days. On day one after an overnight fast, participants reported to the laboratory and were presented with 11, 5 gram portions of almonds to chew 10, 25, or 40 times, depending on treatment arm. The participant remained in the laboratory for 4 hours post-almond consumption for measurements of blood and appetite. For the remainder of the 4 days, participants consumed all meals in the laboratory and collected all stools passed. On a separate occasion, recovered particle sizes of masticated almonds were measured by a mechanical sieving process. Individuals chewed almond samples either 10, 25 or 40 times and expectorated them into sieves.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* BMI 20-25 kg/m2
* Full set of healthy teeth
* Weight stable (<3 kg change in past 3 mo)

Exclusion Criteria:

* Smoker
* Eating Disorders or high level of restraint
* Endocrine disorders
* Pregnant or lactating
* Allergic to nuts
* Taking medication likely to confound study outcomes (meds affecting appetite)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University and community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Lipid available for absorption as measured by stool collections, appetite measures, blood analysis | 3, 4 day periods

SECONDARY OUTCOMES:
Particle size distribution as measured by mechanical sieving process | 3 separate sessions

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, MPH, PhD, RD, Principal Investigator — Purdue University; Bridget A Cassady, B.S., Study Director — Purdue University
Locations (1):
- Purdue University, Laboratory forSensory and Ingestive Studies, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Cassady BA, Hollis JH, Fulford AD, Considine RV, Mattes RD. Mastication of almonds: effects of lipid bioaccessibility, appetite, and hormone response. Am J Clin Nutr. 2009 Mar;89(3):794-800. doi: 10.3945/ajcn.2008.26669. Epub 2009 Jan 14. PMID 19144727